CLINICAL TRIAL: NCT00631410
Title: Phase I Study Of Sunitinib In Combination With Oxaliplatin, L-Leucovorin, And 5-Fluorouracil In Patients With Metastatic Colorectal Cancer
Brief Title: Study Of Sunitinib In Combination With Folfox In Patients With Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181148
Record Dates: First submitted 2008-01-02; First posted 2008-03-07 (Estimated); Results first posted 2010-08-17 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Neoplasms
Keywords: Phase 1; CRC; SU011248; Sunitinib; FOLFOX; Colorectal cancer; metastatic carcinoma of the colon or rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: sunitinib + mFOLFOX6
- B (Experimental)
  Interventions: Drug: sunitinib + mFOLFOX6

INTERVENTIONS:
Drug: sunitinib + mFOLFOX6 — 37.5 mg/day, oral, administered on an outpatient basis for 4 weeks on, 2 weeks off (Schedule 4/2)
  Arms: A
Drug: sunitinib + mFOLFOX6 — 50 mg/day, oral, administered on an outpatient basis for 2 weeks on, 2 weeks off (Schedule 2/2)
  Arms: B

SUMMARY:
To assess the safety and tolerability of sunitinib when administered in combination with modified FOLFOX6 in Japanese patients with metastatic colorectal cancer in the first-line treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum with documented locally advanced or metastatic disease.
* Evidence of unidimensionally measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Prior treatment with systemic therapy for locally advanced or metastatic colorectal cancer.
* Prior surgery or investigational agent within 4 weeks prior to study entry.
* Pregnancy or breastfeeding. All female patients of reproductive potential must have a negative pregnancy test (serum or urine) prior to the start of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Japan (3):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Suntougun, Shizuoka
  - Pfizer Investigational Site, Chuo-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181148&StudyName=Study%20Of%20Sunitinib%20In%20Combination%20With%20Folfox%20In%20Patients%20With%20Colorectal%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm A 37.5 mg/Day (4/2): Sunitinib was administered orally in a 4 weeks on, 2 weeks off intermittent dosing regimen, at a starting dose of 37.5 mg/day (37.5 mg/day in Schedule 4/2). A combination chemotherapy of fluorouracil, calcium folinate and oxaliplatin (FOLFOX) was administered on an every-2-week cycle using the mFOLFOX6 regimen consisting of oxaliplatin 85 mg/meter^2 and l-leucovorin 200 mg/meter^2 as a 2-hour intravenous infusion followed by an intravenous bolus of fluorouracil 400 mg/meter^2 and a 46-hour intravenous infusion of fluorouracil 2,400 mg/meter^2 on Days 1 and 2 of each cycle.
- Treatment Arm B 50 mg/Day (2/2): Sunitinib was administered orally in a 2 weeks on, 2 weeks off intermittent dosing regimen, at a starting dose of 50 mg/day (50 mg/day in Schedule 2/2). A combination chemotherapy of fluorouracil, calcium folinate and oxaliplatin (FOLFOX) was administered on an every-2-week cycle using the mFOLFOX6 regimen consisting of oxaliplatin 85 mg/meter^2 and l-leucovorin 200 mg/meter^2 as a 2-hour intravenous infusion followed by an intravenous bolus of fluorouracil 400 mg/meter^2 and a 46-hour intravenous infusion of fluorouracil 2,400 mg/meter^2 on Days 1 and 2 of each cycle.
Period: Overall Study
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2)
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 3
Not completed — Objective Progression or Relapse | 4 | 3
Not completed — Surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm A 37.5 mg/Day (4/2): Sunitinib was administered orally in a 4 weeks on, 2 weeks off intermittent dosing regimen, at a starting dose of 37.5 mg/day (37.5 mg/day in Schedule 4/2). FOLFOX was administered on an every-2-week cycle using the mFOLFOX6 regimen consisting of oxaliplatin 85 mg/meter^2 and l-leucovorin 200 mg/meter^2 as a 2-hour intravenous infusion followed by an intravenous bolus of fluorouracil 400 mg/meter^2 and a 46-hour intravenous infusion of fluorouracil 2,400 mg/meter^2 on Days 1 and 2 of each cycle.
- Treatment Arm B 50 mg/Day (2/2): Sunitinib was administered orally in a 2 weeks on, 2 weeks off intermittent dosing regimen, at a starting dose of 50 mg/day (50 mg/day in Schedule 2/2).
  FOLFOX was administered on an every-2-week cycle using the mFOLFOX6 regimen consisting of oxaliplatin 85 mg/meter^2 and l-leucovorin 200 mg/meter^2 as a 2-hour intravenous infusion followed by an intravenous bolus of fluorouracil 400 mg/meter^2 and a 46-hour intravenous infusion of fluorouracil 2,400 mg/meter^2 on Days 1 and 2 of each cycle.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Number; unit: participants]
  20-44 years | 0 | 0 | 0
  45-64 years | 4 | 3 | 7
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Score 0: Fully active, able to carry on all pre-disease performance without restriction; Score
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as light house work and office work.
  participants
    Score 0 | 5 | 6 | 11
    Score 1 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, adverse events graded as Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE) Grade 3 or higher , serious adverse events, adverse events resulted in discontinuation, treatment interruption, or dose reduction.
Time Frame: Up to 733 days (the last subject study discontinuation)
Population: All subjects who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Groups:
- Treatment Arm A 37.5 mg/Day (4/2): Sunitinib was administered orally in a 4 weeks on, 2 weeks off intermittent dosing regimen, at a starting dose of 37.5 mg/day (37.5 mg/day in Schedule 4/2). FOLFOX was administered on an every-2-week cycle using the mFOLFOX6 regimen consisting of oxaliplatin 85 mg/meter^2 and ℓ-leucovorin 200 mg/meter^2 as a 2-hour intravenous infusion followed by an intravenous bolus of fluorouracil 400 mg/meter^2 and a 46-hour intravenous infusion of fluorouracil 2,400 mg/meter^2 on Days 1 and 2 of each cycle.
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 6 | 6
participants
  Any adverse events | 6 | 6
  Any serious adverse evets | 2 | 4
  Any Grade-3 or -4 adverse evets | 6 | 6
  Any Grade-5 adverse events (= death) | 0 | 0
  Discontinuation due to adverse events | 1 | 3
  Sunitinib interruption due to adverse events | 6 | 6
  mFOLFOX6 interruption due to adverse events | 6 | 6
  Sunitinib dose reduction due to adverse events | 1 | 1
  mFOLFOX6 dose reduction due to adverse events | 2 | 4

2. Secondary Outcome: Plasma Concentration of Sunitinib
Description: Concentrations after administration of sunitinib alone (Day 14 of Cycle 1) and those after administration of sunitinib in combination with mFOLFOX6 (Day 1 of Cycle 2) were evaluated.
Time Frame: Cycle 1 Day 14 and Cycle 2 Day 1
Population: Pharmacokinetic analysis population consisted of subjects with at least 1 plasma drug concentration measurement in the Treatment Arm B.
Measure: Median (Full Range); unit: nanogram per milliliter
Arm/Group | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 4
nanogram per milliliter
  Cycle 1 Day 14, 0 hour post dose | 85.40 [59.7 to 102]
  Cycle 1 Day 14, 2 hour post dose | 86.15 [66.7 to 107]
  Cycle 1 Day 14, 6 hour post dose | 93.35 [86.8 to 101]
  Cycle 1 Day 14, 8 hour post dose | 98.50 [83.8 to 107]
  Cycle 2 Day 1, 0 hour post dose | 81.70 [71.3 to 97.9]
  Cycle 2 Day 1, 2 hour post dose | 87.05 [81.3 to 90.9]
  Cycle 2 Day 1, 6 hour post dose | 109.50 [102 to 115]
  Cycle 2 Day 1, 8 hour post dose | 102.00 [92.8 to 116]
  Cycle 2 Day 1, 24 hour post dose | 81.50 [79.3 to 96.1]

3. Secondary Outcome: Plasma Concentration of Sunitinib Active Metabolite (SU012662)
Description: as for outcome 2
Time Frame: Cycle 1 Day 14 and Cycle 2 Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: nanogram per milliliter
Arm/Group | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 4
nanogram per milliliter
  Cycle 1 Day 14, 0 hour post dose | 41.75 [16.1 to 59.2]
  Cycle 1 Day 14, 2 hour post dose | 36.90 [18.4 to 68.5]
  Cycle 1 Day 14, 6 hour post dose | 43.55 [19.8 to 58.9]
  Cycle 1 Day 14, 8 hour post dose | 42.35 [18.8 to 64.9]
  Cycle 2 Day 1, 0 hour post dose | 42.65 [19.6 to 62.4]
  Cycle 2 Day 1, 2 hour post dose | 36.10 [23.4 to 61.2]
  Cycle 2 Day 1, 6 hour post dose | 46.95 [23.4 to 67]
  Cycle 2 Day 1, 8 hour post dose | 47.10 [25.7 to 70.1]
  Cycle 2 Day 1, 24 hour post dose | 44.85 [21.7 to 60.5]

4. Secondary Outcome: Plasma Concentration of the Total Drug (Sunitinib Plus SU012662)
Description: as for outcome 2
Time Frame: Cycle 1 Day 14 and Cycle 2 Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: nanogram per milliliter
Arm/Group | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 4
nanogram per milliliter
  Cycle 1 Day 14, 0 hour post dose | 136.25 [75.8 to 143]
  Cycle 1 Day 14, 2 hour post dose | 123.05 [85.1 to 175.5]
  Cycle 1 Day 14, 6 hour post dose | 136.75 [106.9 to 159.9]
  Cycle 1 Day 14, 8 hour post dose | 142.35 [102.6 to 168.9]
  Cycle 2 Day 1, 0 hour post dose | 132.85 [90.9 to 143.3]
  Cycle 2 Day 1, 2 hour post dose | 122.15 [114.3 to 144.5]
  Cycle 2 Day 1, 6 hour post dose | 155.45 [133.4 to 176]
  Cycle 2 Day 1, 8 hour post dose | 156.60 [118.5 to 171.1]
  Cycle 2 Day 1, 24 hour post dose | 132.15 [101.7 to 144.3]

5. Secondary Outcome: Best Overall Response Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Complete response (CR): 2 or more sequential occasions of documented objective disappearance of all target lesions at a minimum of 4 weeks apart; partial response (PR): 2 or more occasions of >=30% decrease in the sum of the longest diameter (LD) of the target lesions from baseline at a minimum of 4 weeks apart; stable disease (SD): at least 1 objective status of stable/no response at least 6 weeks after enrollment; progressive disease (PD): Objective status of progression within 12 weeks of enrollment, not qualifying as CR, PR or Stable; Indeterminate: no other response category applies.
Time Frame: Up to the last subject completed Cycle 24 or individual study discontinuation
Population: All enrolled subjects who 1) had a diagnosis of locally-advanced or metastatic adenocarcinoma of the colon or rectum with measurable disease at baseline; 2) had received at least one dose of the investigational product; and 3) with efficacy data available after administration of the investigational product.
Measure: Number; unit: participants
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 6 | 6
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 4 | 4
  Stable Disease (SD) | 1 | 1
  Progressive Disease (PD) | 1 | 0
  Indeterminate | 0 | 1
  Objective Response (CR+PR) | 4 | 4

6. Secondary Outcome: Duration of Response (DR)
Description: Duration of response is defined as the duration from the date of first documentation of complete response (CR) or partial response (PR) to date of first documentation of objective progression based on the investigator's assessment.
Time Frame: Up to 733 days (the last subject study discontinuation)
Population: Summary statistics were not calculated due to a small number of subjects.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the time from date of enrolment to date of first documentation of progression based on investigator's assessment or death due to any cause.
Time Frame: Up to 733 days (the last subject study discontinuation)
Population: Summary statistics were not calculated due to a small number of subjects.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Sunitinib Relative Dose Intensity in the Treatment Arm A
Description: Relative dose intensity is defined as percentage of total dose administered over total dose assigned through assessment period. Period 1: Cycle 1 to 3; Period 2: Cycle 4 to 6; Period"n": Cycle (n-1)*3+1 to n*3.
Time Frame: Up to 733 days (the last subject study discontinuation in the Treatment Arm A)
Population: All subjects who received at least 1 dose of the study drug. n = number of subjects assessed for relative dose intensity in the given period.
Measure: Mean (Standard Deviation); unit: percent of total planned dose
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2)
Number analyzed (Participants) | 6
percent of total planned dose
  Period 1 (n=6) | 57.1 (9.3)
  Period 2 (n=5) | 72.4 (18.5)
  Period 3 (n=5) | 64.3 (21.1)
  Period 4 (n=4) | 53.6 (15.4)
  Period 5 (n=3) | 42.9 (16.5)
  Period 6 (n=2) | 50.0 (0.0)
  Period 7 (n=2) | 40.5 (37.0)
  Period 8 (n=1) | 50.0 (0)
  Period 9 (n=1) | 50.0 (0)
  Period 10 (n=1) | 23.8 (0)
  Period 11 (n=1) | 33.3 (0)
  Period 12 (n=1) | 23.8 (0)
  Period 13 (n=1) | 25.0 (0)
  Period 14 (n=1) | 33.3 (0)
  Period 15 (n=1) | 23.8 (0)
  Period 16 (n=1) | 25.0 (0)

9. Secondary Outcome: Sunitinib Relative Dose Intensity in the Treatment Arm B
Description: Relative dose intensity is defined as percentage of total dose administered over total dose assigned through assessment period. Period 1: Cycle 1 to 2; Period 2: Cycle 3 to 4, Period"n": Cycle (n-1)*2+1 to n*2.
Time Frame: Up to 384 days (the last subject study discontinuation in the Treatment Arm B)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent of total planned dose
Arm/Group | Treatment Arm B 50 mg/Day (2/2)
Number analyzed (Participants) | 6
percent of total planned dose
  Period 1 (n=6) | 100.0 (0)
  Period 2 (n=5) | 97.1 (3.9)
  Period 3 (n=5) | 78.6 (23.6)
  Period 4 (n=5) | 90.0 (13.7)
  Period 5 (n=5) | 82.1 (11.0)
  Period 6 (n=3) | 73.8 (26.8)
  Period 7 (n=3) | 75.0 (25.0)
  Period 8 (n=3) | 75.0 (25.0)
  Period 9 (n=3) | 73.8 (26.8)
  Period 10 (n=3) | 73.8 (26.8)
  Period 11 (n=1) | 100.0 (0)
  Period 12 (n=1) | 35.7 (0)

ADVERSE EVENTS:
Time Frame: Up to 733 days (the last subject study discontinuation)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Treatment Arm A 37.5 mg/Day (4/2) | Treatment Arm B 50 mg/Day (2/2)
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm A 37.5 mg/Day (4/2) (N=6) | Treatment Arm B 50 mg/Day (2/2) (N=6)
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm A 37.5 mg/Day (4/2) (N=6) | Treatment Arm B 50 mg/Day (2/2) (N=6)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Thyroid disorder (Endocrine disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 5 | 3
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 5 | 5
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood albumin decreased (Investigations) | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Blood amylase increased (Investigations) | 2 | 2
Blood calcium decreased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 3
Blood phosphorus increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 2 | 0
Blood sodium decreased (Investigations) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 3
Blood urea increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Glucose urine (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 3 | 5
Lymphocyte count decreased (Investigations) | 3 | 5
Neutrophil count decreased (Investigations) | 6 | 6
Platelet count decreased (Investigations) | 6 | 6
Protein total decreased (Investigations) | 1 | 0
Protein urine (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 6 | 6
Anorexia (Metabolism and nutrition disorders) | 5 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Neurotoxicity (Nervous system disorders) | 0 | 4
Parosmia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 2 | 3
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Implant site haematoma (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.